CLINICAL TRIAL: NCT05243381
Title: Inflammation, NK Cells, Antisense Protein and Exosomes, and Correlation With Immune Response During HIV Infection
Acronym: INKASE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RECHMPL21_0518
Record Dates: First submitted 2022-01-24; First posted 2022-02-17 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: HIV Infections
Keywords: Immune non-responder HIV-patients; Immune responder HIV-patients; HIV-1 antisense protein; Exosomes; NK cells
MeSH Terms: conditions — HIV Infections | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immune non-responder patients (Other): * HIV viral load < 50 copies/ml in the past 2 years
  * CD4+ T-cell count < 350 cells/mm3 on the last two tests
  Interventions: Biological: 20 ml blood test
- Immune responder patients (Other): * HIV viral load < 50 copies/ml in the past 2 years
  * CD4+ T-cell count > 500 cells/mm3 on the last two tests
  Interventions: Biological: 20 ml blood test

INTERVENTIONS:
Biological: 20 ml blood test — 20 ml blood test

SUMMARY:
More than 90% of HIV-infected patients on antiretroviral therapy have an undetectable viral load. However, approximately 15% of these individuals do not sufficiently restore their TCD4 lymphocytes and have an unfavorable CD4/CD8 ratio despite good adherence and an undetectable viral load. Factors associated with immunovirological discordance include low CD4 cell counts prior to antiretroviral therapy, low CD4/CD8 ratios and positive cytomegalovirus (CMV) serology. These patients are at risk of significant non-AIDS events and mortality.

The anti-sense protein (ASP) is synthesized from the anti-sense strand of HIV-1. A cytotoxic anti-ASP response of CD8 T lymphocytes and anti-ASP antibodies have been demonstrated in infected patients. The conservation of the ASP gene in HIV-1, the virus responsible for the pandemic, suggests that its maintenance confers an advantage to the virus. ASP induces an inflammatory phenotype in surrounding cells. ASP can be externalized by the cell through its interaction with its cellular partner Bat-3. Once externalized in soluble or exosomal form, Bat-3 has the ability to regulate NK cell activity. During HIV infection, NK functions are disrupted, including those related to the expression of the Bat-3 receptor, NKp30.

In patients, the inflammatory phenomenon is strongly associated with chronic HIV-1 infection. The efficacy of antiviral treatments does not allow a complete normalization of either the immune system function or the inflammatory status of the patient. The observed effect of ASP on inflammation raises the question of the involvement of ASP in the maintenance of a chronic inflammatory state in patients under treatment. Increased inflammation has also been associated in HIV-infected patients with elevated plasma exosome levels. In patients undergoing treatment, chronic inflammation remains a major problem and an important source of comorbidities (cardiovascular in particular) and probably contributes to the immunovirological non-response in immunodiscordant HIV-infected patients.

It is hypothesized that ASP bound to its cellular partner Bat-3 in exosomes would disrupt the cytotoxic activity of NK cells, sustain inflammation and have a deleterious effect on immune reconstitution.

DETAILED DESCRIPTION:
The main objective of the project is to characterize the presence of ex vivo NK cell perturbations in patients living with HIV (PLHIV) with immunovirological discordance, in relation to ASP expression and plasmatic exosomes. The secondary objectives will be to identify new biological parameters to study and to establish mechanistic hypothesis explaining the results obtained during the study.

The study has a pathophysiological aim and is approved by the committee for the protection of individuals. Two groups of patients will be constituted: one group of PLWHIV with immunovirological discordance (20 patients) and the other group of PLWHIV with a good immune reconstitution (40 patients).

ELIGIBILITY:
Inclusion Criteria:

* Patiens living with HIV over 45 years old
* At least 2 measurements of CD4+ T-cell and HIV viral load in the last 2 years
* HIV viral load < 50 copies/ml in the past 2 years
* For the immune non-responder patients : CD4+ T-cell count < 350 cells/mm3 on the last two tests
* For the immune responder patients: CD4+ T-cell count > 500 cells/mm3 on the last two tests

Exclusion Criteria:

* No antiretroviral treatment
* Immunosuppressive treatment
* History of cancer less than 5 years
* Pregnancy
* Breastfeeding mother
* Adult protected by law or patient under guardianship or curatorship
* Failure to obtain written informed consent after a reflection period
* Not be affiliated to a French social security system or a beneficiary of such a system

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-04-22 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Immune status of HIV-infected patients | The day of inclusion
  CD4+ T-cell count

SECONDARY OUTCOMES:
HIV-1 Antisense protein | The day of inclusion
  HIV-1 antisense protein expression level
Impacts of exosomes on NK cell activity | The day of inclusion
  Cytotoxicity activity and cytokines production (intracellular staining and qRT-PCR) during cytotoxicity assay
NK cells phenotyping | The day of inclusion
  Flow cytometry phenotyping: subpopulation, activation and exhaustion markers
NK cells functionality | The day of inclusion
  Natural and antibody-dependent cytotoxicity assays

CONTACTS AND LOCATIONS:
Overall Officials: Alain MAKINSON, MH PD, Principal Investigator — UH MONTPELLIER; Antoine GROSS, PHD, Study Director — Centre National de la Recherche Scientifique, France
Locations (1):
- La Colombiere Hospital, Montpellier, Herault, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Landry S, Halin M, Lefort S, Audet B, Vaquero C, Mesnard JM, Barbeau B. Detection, characterization and regulation of antisense transcripts in HIV-1. Retrovirology. 2007 Oct 2;4:71. doi: 10.1186/1742-4690-4-71. PMID 17910760
- [Background] Laverdure S, Gross A, Arpin-Andre C, Clerc I, Beaumelle B, Barbeau B, Mesnard JM. HIV-1 antisense transcription is preferentially activated in primary monocyte-derived cells. J Virol. 2012 Dec;86(24):13785-9. doi: 10.1128/JVI.01723-12. Epub 2012 Oct 3. PMID 23035216
- [Background] Bet A, Maze EA, Bansal A, Sterrett S, Gross A, Graff-Dubois S, Samri A, Guihot A, Katlama C, Theodorou I, Mesnard JM, Moris A, Goepfert PA, Cardinaud S. The HIV-1 antisense protein (ASP) induces CD8 T cell responses during chronic infection. Retrovirology. 2015 Feb 10;12:15. doi: 10.1186/s12977-015-0135-y. PMID 25809376
- [Background] Savoret J, Chazal N, Moles JP, Tuaillon E, Boufassa F, Meyer L, Lecuroux C, Lambotte O, Van De Perre P, Mesnard JM, Gross A. A Pilot Study of the Humoral Response Against the AntiSense Protein (ASP) in HIV-1-Infected Patients. Front Microbiol. 2020 Jan 24;11:20. doi: 10.3389/fmicb.2020.00020. eCollection 2020. PMID 32117090
- [Background] Cassan E, Arigon-Chifolleau AM, Mesnard JM, Gross A, Gascuel O. Concomitant emergence of the antisense protein gene of HIV-1 and of the pandemic. Proc Natl Acad Sci U S A. 2016 Oct 11;113(41):11537-11542. doi: 10.1073/pnas.1605739113. Epub 2016 Sep 28. PMID 27681623
- [Background] Wang Y, Lifshitz L, Gellatly K, Vinton CL, Busman-Sahay K, McCauley S, Vangala P, Kim K, Derr A, Jaiswal S, Kucukural A, McDonel P, Hunt PW, Greenough T, Houghton J, Somsouk M, Estes JD, Brenchley JM, Garber M, Deeks SG, Luban J. HIV-1-induced cytokines deplete homeostatic innate lymphoid cells and expand TCF7-dependent memory NK cells. Nat Immunol. 2020 Mar;21(3):274-286. doi: 10.1038/s41590-020-0593-9. Epub 2020 Feb 17. PMID 32066947
- [Background] Giuliani E, Vassena L, Di Cesare S, Malagnino V, Desimio MG, Andreoni M, Barnaba V, Doria M. NK cells of HIV-1-infected patients with poor CD4+ T-cell reconstitution despite suppressive HAART show reduced IFN-gamma production and high frequency of autoreactive CD56bright cells. Immunol Lett. 2017 Oct;190:185-193. doi: 10.1016/j.imlet.2017.08.014. Epub 2017 Aug 19. PMID 28826739
- [Background] Florez-Alvarez L, Hernandez JC, Zapata W. NK Cells in HIV-1 Infection: From Basic Science to Vaccine Strategies. Front Immunol. 2018 Oct 17;9:2290. doi: 10.3389/fimmu.2018.02290. eCollection 2018. PMID 30386329
- [Background] Lucar O, Reeves RK, Jost S. A Natural Impact: NK Cells at the Intersection of Cancer and HIV Disease. Front Immunol. 2019 Aug 14;10:1850. doi: 10.3389/fimmu.2019.01850. eCollection 2019. PMID 31474977
- [Background] Perez PS, Romaniuk MA, Duette GA, Zhao Z, Huang Y, Martin-Jaular L, Witwer KW, Thery C, Ostrowski M. Extracellular vesicles and chronic inflammation during HIV infection. J Extracell Vesicles. 2019 Nov 6;8(1):1687275. doi: 10.1080/20013078.2019.1687275. eCollection 2019. PMID 31998449
- [Background] Pantazis N, Papastamopoulos V, Paparizos V, Metallidis S, Adamis G, Antoniadou A, Psichogiou M, Chini M, Sambatakou H, Sipsas NV, Gogos C, Chrysos G, Panagopoulos P, Katsarou O, Gikas A, Touloumi G; AMACS. Long-term evolution of CD4+ cell count in patients under combined antiretroviral therapy. AIDS. 2019 Aug 1;33(10):1645-1655. doi: 10.1097/QAD.0000000000002248. PMID 31305332
- [Background] Gras L, May M, Ryder LP, Trickey A, Helleberg M, Obel N, Thiebaut R, Guest J, Gill J, Crane H, Dias Lima V, d'Arminio Monforte A, Sterling TR, Miro J, Moreno S, Stephan C, Smith C, Tate J, Shepherd L, Saag M, Rieger A, Gillor D, Cavassini M, Montero M, Ingle SM, Reiss P, Costagliola D, Wit FWNM, Sterne J, de Wolf F, Geskus R; Antiretroviral Therapy Cohort Collaboration (ART-CC). Determinants of Restoration of CD4 and CD8 Cell Counts and Their Ratio in HIV-1-Positive Individuals With Sustained Virological Suppression on Antiretroviral Therapy. J Acquir Immune Defic Syndr. 2019 Mar 1;80(3):292-300. doi: 10.1097/QAI.0000000000001913. PMID 30531492
- [Background] Roul H, Mary-Krause M, Ghosn J, Delaugerre C, Pialoux G, Cuzin L, Launay O, Lacombe JM, Menard A, De Truchis P, Delfraissy JF, Weiss L, Costagliola D; FHDH-ANRS CO4. CD4+ cell count recovery after combined antiretroviral therapy in the modern combined antiretroviral therapy era. AIDS. 2018 Nov 13;32(17):2605-2614. doi: 10.1097/QAD.0000000000002010. PMID 30289817
- [Background] Mussini C, Lorenzini P, Cozzi-Lepri A, Lapadula G, Marchetti G, Nicastri E, Cingolani A, Lichtner M, Antinori A, Gori A, d'Arminio Monforte A; Icona Foundation Study Group. CD4/CD8 ratio normalisation and non-AIDS-related events in individuals with HIV who achieve viral load suppression with antiretroviral therapy: an observational cohort study. Lancet HIV. 2015 Mar;2(3):e98-106. doi: 10.1016/S2352-3018(15)00006-5. Epub 2015 Feb 6. PMID 26424550